CLINICAL TRIAL: NCT05755685
Title: Hyperthermic Intraperitoneal Treatment of Recombinant Modified Human Tumor Necrosis Factor (rmhTNF) for Colorectal Cancer With Peritoneal Metastases: Phase II Clinical Trial
Brief Title: Hyperthermic Intraperitoneal Treatment of rmhTNF for CRCPM: Phase II Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai Weike Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-0966
Record Dates: First submitted 2023-02-07; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Peritoneal Metastases; Colorectal Cancer
Keywords: Colorectal Cancer; Peritoneal metastasis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group1 (Experimental): The preoperative clinical stage was M1c colon or peritoneal retroflex superior rectum adenocarcinoma
  Interventions: Drug: Hyperthermic intraperitoneal treatment of recombinant modified human tumor necrosis factor (rmhTNF)

INTERVENTIONS:
Drug: Hyperthermic intraperitoneal treatment of recombinant modified human tumor necrosis factor (rmhTNF) — 5 million IUrmhTNF, dissolved in 30-50ml normal saline, was intraperitoneal heat perfusion into the surgical focus after the operation;

SUMMARY:
The goal of this study is planing to adopt intra-abdominal perfusion therapy of rmhTNF during radical colorectal cancer surgery to determine whether intra-abdominal therapy has an impact on postoperative intestinal function recovery, anastomotic leakage, postoperative bleeding, postoperative adhesion intestinal obstruction and other complications. On this basis, the effect of rmhTNF on postoperative peritoneal implantation metastasis and long-term survival was further studied. The main question it aims to answer is: To evaluate the safety and efficacy of rmhTNF in the treatment of peritoneal metastases in colorectal cancer. Participants will receive 1. Radical surgery: Surgical methods can be developed or endoscopic (including robotic surgery). Radical resection of colorectal cancer (corresponding resection of colon and rectum plus regional lymph node dissection, regional lymph node dissection including parenteral, intermediate and mesangial root lymph nodes) follows the principle of mesangectomy and tumorless operation. 2. Abdominal heat perfusion was performed twice: the first time, 5 million IUrmhTNF, dissolved in 30-50ml normal saline, was intraperitoneal heat perfusion into the surgical focus after the operation; the second time, rhatitrexed 2.5mg/m2 was injected into the abdominal cavity through thermoperfusion or drainage tube; 3. Postoperative systemic chemotherapy regimen: postoperative adjuvant chemotherapy should be started 3-4 weeks after surgery, and appropriately extended for patients with poor physique, but no later than 8 weeks after surgery. The chemotherapy regimen was determined by the clinician according to pathological stage, molecular typing, and risk factors, referring to the NCCN and CSCO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of colonic and peritoneal reflexive superior rectum was confirmed by pathology, aged 18-70 years;
* Body condition score (PS) 0 ~ 1 in the Eastern Tumor Collaboration Group (ECOG);
* Preoperative clinical stage was M1c;
* No neoadjuvant therapy was performed;
* Histopathologically confirmed as peritoneal metastases of colorectal cancer > 10cm from the anus, R0-resected, adenocarcinoma/mucinous adenocarcinoma
* The functions of vital organs shall meet the following requirements;
* Be able to understand the situation of this study and sign informed consent.

Exclusion Criteria:

* Allergic history of TNF and its derivatives;
* Patients with fever (>38℃);
* Active hepatitis and peripheral neuropathy (e.g., peripheral neuritis, pseudomeningitis, motor neuritis, and sensory disorders);
* Pregnant or lactating women, or potentially pregnant women and sexually active men who refuse/cannot receive medically acceptable forms of contraception;
* Patients with a history of malignant tumor;
* Clinical symptoms or diseases of the heart that are not well controlled.
* Subject has any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism;
* The subject has a known history of psychotropic substance abuse, alcoholism or drug use; Subjects innate or acquired immune function defects (such as HIV infection), or active hepatitis
* Other conditions in which the investigator thinks the patient should not participate in the study;
* A history of neurological or psychiatric disorders, such as major depression or dementia, that may affect the informed study or follow-up evaluation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, the time of postoperative intestinal function recovery, whether exist anastomotic leakage, postoperative bleeding, postoperative adhesion ileus, and other complications in 2 weeks after surgery.

SECONDARY OUTCOMES:
the recurrence rate of metastasis and long-term survival of participants accepted the treatment of rmhTNF in the treatment of peritoneal metastases in colorectal cancer. | 1 year
  1. record the time period between the date of randomization and the date of patient tumor recurrence or death (earliest occurrence), and calculated the recurrence rate of metastasis after surgery.
  2. 1-year overall survival rate after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lifeng Sun, Dr, Study Chair — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China